CLINICAL TRIAL: NCT06227871
Title: A Retrospective Analysis of Pancreatic Injuries and Treatment Outcomes
Status: Completed | Type: Observational
Sponsor: Kern Medical Center (Other)
Responsible Party: Principal Investigator, Amber Jones, Principal Investigator, DO, MPH, Kern Medical Center
Other Study IDs: 11894
Record Dates: First submitted 2024-01-17; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Trauma; Pancreatic Duct Injury; Pancreas Necrosis; Pancreas Cyst; Pancreas; Fistula; Pancreas Abscess; Intra-Abdominal Abscess; Anastomotic Leak; Pancreas Injury
Keywords: Pancreatic trauma; Penetrating abdominal injury; Abdominal trauma
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatic Cyst; Pancreatic Fistula; Abdominal Abscess; Anastomotic Leak; Abdominal Injuries | interventions — Laparotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Penetrating intra-abdominal injury: Patients diagnosed with a pancreatic injury secondary to penetrating intra-abdominal injury subdivided by pancreatic injury grade
  Interventions: Procedure: Exploratory laparotomy
- Blunt intra-abdominal injury: Patients diagnosed with a pancreatic injury secondary to blunt intra-abdominal injury subdivided by pancreatic injury grade
  Interventions: Procedure: Exploratory laparotomy

INTERVENTIONS:
Procedure: Exploratory laparotomy — Exploratory laparotomy with interventions addressing pancreatic injuries Grade 1-5 including pancreatic interventions including subtotal pancreatectomy, distal pancreatectomy, pancreatic ligation, pyloric diversion, or simple drainage of the pancreas.

SUMMARY:
The goal of this observational study is to compare the presentation, treatment, and outcomes in patients suffering traumatic pancreatic injuries from blunt or penetrating trauma.

The questions this study aims to answer are:

1. Does a statistically significant association exist between pancreatic injury grade and the following individual factors:

   * Mortality
   * Morbidity
   * Injury severity score
2. Is there an association between post-operative pancreatic complications and operation-specific intervention?
3. Does pancreatic injury score correlate with certain intra-abdominal organ injuries?

Participants meeting criteria are greater than 18 years old, with no history of pancreatic surgery who were hospitalized at Kern Medical Center after presenting to the institution's emergency department as tier 1 or 2 trauma activations following blunt or penetrating abdominal injury and were diagnosed with pancreatic injury during the same hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized at Kern Medical Center after presenting to the institution's emergency department as a tier 1 and 2 trauma activation
* Hospitalized following blunt or penetrating abdominal injury
* Diagnosed with traumatic pancreatic injury during same admission

Exclusion Criteria:

* history of pancreatic surgery
* Iatrogenic pancreatic injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's greater than 18 years old, with no history of pancreatic surgery who were hospitalized at Kern Medical Center from November 1st, 2019 to March 1st, 2023 after presenting to the institution's emergency department as tier 1 and 2 trauma activations following blunt or penetrating abdominal injury and were diagnosed with pancreatic injury during the same hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Complication occurrence | Up to 12 weeks postoperatively
  Complications including wound dehiscence, pancreatic duct leak, pancreatic pseudocyst, pancreatic fistula formation, pancreatic necrosis, intra-abdominal abscess, traumatic pancreatitis, anastomotic leak

SECONDARY OUTCOMES:
Associated intra-abdominal injuries | within 48 hours of admission
  concomitant intra-abdominal injuries including pancreatic duck, diaphragm, stomach, liver, kidney, Major vasculature, spleen, duodenum, small bowel, colon, ureter

CONTACTS AND LOCATIONS:
Overall Officials: Amber Jones, DO, MPH, Principal Investigator — Kern Medical Center
Locations (1):
- Kern Medical Center, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No